CLINICAL TRIAL: NCT03673098
Title: Developing a Resilience Intervention for Older, HIV-Infected Women
Brief Title: The BRIgHT Program: Building Resilience in HIV Together
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Christina Psaros, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018P001803; 5R34AT009170 (NIH)
Record Dates: First submitted 2018-09-04; First posted 2018-09-17 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Resilience, Psychological
Keywords: Resilience; Women; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Intervention: 10 weekly sessions of the adapted Relaxation Response Resiliency Program (3RP) Control: 10 weekly sessions of a supportive psychotherapy program
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Adapted 3RP (Experimental): The intervention condition will consist of the 10-week adapted 3RP intervention.
  Interventions: Behavioral: Adapted 3RP
- Control Group: Supportive Psychotherapy (No Intervention): The control condition will be a 10-week supportive therapy program. Visits include supportive psychotherapy to address stressful or difficult topics related to aging as a woman living with HIV. The program was developed to approximate the most frequent mental health counseling provided to adults with HIV at the community level.

INTERVENTIONS:
Behavioral: Adapted 3RP — The 3RP blends stress management principles, cognitive behavioral therapy, and positive psychology. The 3RP focuses on 3 major areas: (1) eliciting the relaxation response; (2) increasing stress awareness; and (3) promoting adaptive strategies. The adapted 3RP intervention consists of 10, 90-minute weekly group sessions. Content specific to older women living with HIV, including self-compassion exercises, was added to the intervention in the first phase of this study (open pilot).
  Arms: Intervention Group: Adapted 3RP

SUMMARY:
This is the second phase of a two-part study. In the first phase (Protocol ID: R34AT009170), the investigators refined and piloted the Relaxation Response Resiliency (3RP) intervention for women age 50 and over who are living with HIV, a group especially burdened by stressors related both to aging and to living with chronic disease. In this part of the study, the investigators will use data from the first phase to further adapt the intervention manual, and test the final product via a small randomized controlled trial in the same population.

DETAILED DESCRIPTION:
Overview.

This is the second phase of a two-part study. In the first phase (Protocol ID: R34AT009170), the investigators adapted an existing resiliency intervention, the Relaxation Response Resiliency Program (3RP), to the needs of women ages 50 and over who are living with HIV. The investigators conducted preliminary testing of the refined group intervention via an open pilot study (N=13 enrolled) across two sites, MGH and Boston Medical Center), and conducted individual exit interviews to solicit feedback on the intervention. Based on these qualitative data, as well as qualitative work conducted previously with this population, the goal of this phase of the project is to conduct a small, randomized pilot of the intervention in groups of up to 10 women with HIV (total N=up to 60) to assess feasibility and acceptability of all study procedures.

Study Procedures.

Participants will be women living with HIV (N=up to 60) age 50 or over, who are recruited via flyers and provider referral from Boston area hospitals and health care settings, as well as community organizations serving individuals living with HIV. Once an individual expresses interest in the study, they will be screened by a study staff member, either by phone or in person, in order to assess study eligibility. Eligible and interested individuals will be invited to sign informed consent and complete an in-person baseline assessment. Participants will be randomized to either a 10-week intervention group (adapted 3RP intervention) or a 10-week control group (supportive psychotherapy program). Participants will then complete a post-treatment assessment, an individual in-depth exit interview to provide feedback on their experience in the study, and a 3-month follow-up assessment. Data from this second phase of the study will inform the eventual development of a full-scale randomized controlled trial.

Adapted 3RP Intervention.

Once randomized into the intervention condition, participants will complete 10, 90-minute weekly group sessions of the adapted 3RP intervention. Sessions will focus on developing an understanding of stress sources and physiology, and on developing a regular practice of eliciting the relaxation response (RR) and learning cognitive behavioral and positive psychology skills to enhance resiliency to long-term stress. Participants will be encouraged to practice skills (RR practice, thoughts records to learn adaptive thinking) between group sessions.

Supportive Psychotherapy Control Program.

The control condition will be a supportive therapy program that is matched to the intervention for number and length of sessions. Basic principles of supportive psychotherapy will be followed, and the interventionist will facilitate discussion around what it is like to live with HIV as an aging woman.

ELIGIBILITY:
Inclusion Criteria:

* biologically born women who endorse a female identity
* living with HIV/AIDS
* age 50 or older
* English-speaking

Exclusion Criteria:

* presence of an active (i.e. untreated) and interfering psychiatric disorder (e.g., bipolar disorder, schizophrenia, substance abuse)
* have participated in a structured cognitive behavioral therapy and/or a mind-body intervention in the past year

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators will recruit biologically born women who endorse a female gender identity.
Enrollment: 44 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Christina, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Boston-area hospitals and healthcare settings between October 2018 and July 2020. The first participant was enrolled on November 5, 2018 and the last participant was enrolled in July 10, 2020.
Pre-assignment Details: Of the 65 participants screened, 61 met inclusion criteria, and 44 were consented, enrolled and randomized to either the intervention arm or the control arm.
Period: Overall Study
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy
Started | 23 | 21
Completed | 13 | 17
Not Completed | 10 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Could not participate due to scheduling conflicts or health issues | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Continuous [Mean (Full Range); unit: years] | 57.6 [50 to 73] | 59.2 [50 to 71] | 58 [50 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 10 | 24
  White | 5 | 8 | 13
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44
Education Level [Count of Participants; unit: Participants]
  No formal education | 0 | 0 | 0
  Eighth grade or lower | 3 | 0 | 3
  Some high school | 3 | 3 | 6
  High school graduate or GED | 5 | 9 | 14
  Some college/Associate degree/technical school | 10 | 5 | 15
  College graduate (BA/BS) | 0 | 1 | 1
  Some graduate school | 1 | 1 | 2
  Master's degree | 1 | 1 | 2
  Doctorate/Medical degree/Law degree | 0 | 0 | 0
  Not Reported | 0 | 1 | 1
Employment Status [Count of Participants; unit: Participants]
  Full-time employed | 5 | 4 | 9
  Part-time Employed | 2 | 4 | 6
  Full-time or part-time in school | 0 | 0 | 0
  Neither employed nor in school/ Retired | 8 | 3 | 11
  On disability | 6 | 9 | 15
  Other | 2 | 1 | 3
Annual Income [Count of Participants; unit: Participants]
  $10,000 or less | 5 | 6 | 11
  $10,001 to $20,000 | 9 | 8 | 17
  $20,001 to $40,000 | 3 | 1 | 4
  $40,001 to $60,000 | 3 | 4 | 7
  $60,001 to $80,000 | 0 | 1 | 1
  Over $80,000 | 2 | 1 | 3
  Not Reported | 1 | 0 | 1
Time Since HIV Diagnosis [Mean (Full Range); unit: years] | 25 [4 to 42] | 27 [14 to 36] | 26 [4 to 42]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Study Procedures, as Assessed by Number of Individuals Screened and Eligible for Participation in the Study
Description: Investigators assessed feasibility of study procedures by tracking the number of potential participants screened and eligible for participation. These metrics were assessed together with the number of eligible individuals enrolled, and the number of assessments completed in order to provide a comprehensive understanding of the feasibility of this study.
Time Frame: Assessed at screening (pre-baseline)
Population: 65 total participants were recruited and screened for eligibility. 61 participants were deemed eligible based on inclusion criteria; 4 were ineligible.
Measure: Count of Participants; unit: Participants
Groups:
- Total Recruitment Population: Feasibility was defined a priori, and was considered met if: (1) ≥ 70% of eligible individuals enrolled in the study; (2) ≥ 7 out of 10 group sessions were attended by ≥ 70% of participants; and (3) ≥ 2 assessments were completed by ≥ 70% of participants.
Arm/Group | Total Recruitment Population
Number analyzed (Participants) | 65
Participants
  Eligible | 61
  Ineligible: Not a cisgender woman | 3
  Ineligible: Not living with HIV | 1

2. Primary Outcome: Feasibility of Study Procedures, as Assessed by Number of Individuals Enrolled and Number of Assessments and Sessions Completed by Enrolled Individuals.
Description: Investigators assessed feasibility of study procedures by tracking the number of eligible participants enrolled, and the number of treatment, assessment, and make-up sessions completed by all enrolled participants. These metrics were assessed together with the number of individuals screened and eligible in order to provide a comprehensive understanding of the feasibility of this study.
Time Frame: Assessed up to 6 months post-baseline
Population: Feasibility was defined a priori, and was considered met if: (1) ≥ 70% of eligible individuals enrolled in the study; (2) ≥ 7 out of 10 group sessions were attended by ≥ 70% of participants; and (3) ≥ 2 assessments were completed by ≥ 70% of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy
Number analyzed (Participants) | 23 | 21
Participants
  Participated in group sessions | 20 | 21
  Attended at least 70% of group sessions | 15 | 15
  Completed post-treatment assessment | 16 | 18
  Completed qualitative exit interview | 15 | 18
  Completed 3-month follow-up assessment | 13 | 17
  Completed COVID-19 quantitative assessment | 13 | 15
  Completed COVID-19 qualitative interview | 10 | 14

3. Primary Outcome: Feasibility of Study Procedures, as Assessed by Time Required for Screening and Enrollment
Description: Investigators assessed feasibility of study procedures by tracking the time it takes to screen and enroll participants, as measured by the number of months it took to recruit, screen, and schedule a baseline assessment for all 44 participants, compared to the number of months we estimated it would take to enroll our target number of participants at the outset of the study (11 months). These metrics were assessed in order to provide a comprehensive understanding of the feasibility of this study.
Time Frame: Assessed after completion of all baseline assessments
Population: Enrollment was expected to begin in April 2018 and end in March 2019, but began instead in October 2018 and ended in July 2020. Total target enrollment for Aim 2 was 60 participants. A total of 65 individuals were screened, 61 were eligible, and 44 were consented/enrolled.
Measure: Number; unit: months
Groups:
- Overall: Total participants (includes both control and intervention)
Arm/Group | Overall
Number analyzed (Participants) | 44
months
  Planned duration of screening and enrollment | 11
  Actual duration of screening and enrollment | 21

4. Primary Outcome: Feasibility of Study Procedures, as Assessed by Time Required to Complete Study Procedures
Description: Investigators assessed feasibility of study procedures by tracking the time it takes for participants to complete each assessment. These metrics were assessed in order to provide a comprehensive understanding of the feasibility of this study.
Time Frame: Assessed up to 6 months post-baseline
Population: Note: Not at all participants in the study completed all time point assessments and/or qualitative interviews. Average time taken to complete the following assessments is based on the specific number of individuals that completed the specific time point assessment rather than the total number of participants enrolled (N=44).
Measure: Mean (Full Range); unit: minutes
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy | Overall
Number analyzed (Participants) | 23 | 21 | 44
minutes
  Baseline assessment | 94.9 [36 to 203] | 94.6 [39 to 184] | 94.8 [36 to 203]
  Post-treatment assessment: number analyzed (Participants) | 16 | 18 | 34
  Post-treatment assessment | 86.7 [33 to 165] | 84.3 [33 to 160] | 85.4 [33 to 165]
  3-month follow-up assessment: number analyzed (Participants) | 13 | 17 | 30
  3-month follow-up assessment | 93.2 [45 to 278] | 70.3 [29 to 138] | 80.9 [29 to 278]

5. Primary Outcome: Feasibility as Assessed by Reasons for Declining Enrollment
Description: Includes the number of individuals who were eligible (N=61), but declined to enroll and those reasons for declining.
Time Frame: Assessed at screening (pre-baseline)
Population: 65 total participants were recruited and screened for eligibility at the outset of the study. 61 were deemed eligible to participate prior to randomization.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Total participants eligible, but declined to enroll.
Arm/Group | Overall
Number analyzed (Participants) | 17
Participants
  Scheduling conflicts | 2
  Lack of interest | 1
  Reason unknown | 14

6. Primary Outcome: Feasibility as Assessed by Reasons for Enrolling But Not Taking Part in Group Sessions
Description: Includes the number of individuals who enrolled, but did not take part in group sessions (N=2) and the reasons for not participating.
Time Frame: Assessed up to 3 months post-baseline
Population: Participants who enrolled but did not attend group sessions (n=2) were part of the intervention arm only (n=2); no participants who enrolled but did not attend group sessions were part of the control arm (n=0). Therefore, the "Overall Number of Participants Analyzed" below are 2 and 0 for the intervention and control arms, respectively, with reasons defined for not taking part in group sessions.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Total participants that enrolled, but did not take part in the group sessions.
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy | Overall
Number analyzed (Participants) | 2 | 0 | 2
Participants
  Scheduling conflicts | 1 | 0 | 1
  Health issues | 1 | 0 | 1

7. Primary Outcome: Feasibility as Assessed by Reasons for Withdrawing From the Study
Description: Includes the number of individuals who withdrew from the study, despite participating in group sessions (N=7), and the reasons for withdrawing.
Time Frame: Assessed up to 6 months post-baseline
Population: Participants who withdrew from the study (n=7) were part of both the intervention arm (n=6) and the control arm (n=1). Therefore, the "Overall Number of Participants Analyzed" below are 6 and 1 for the intervention and control arms, respectively, with reasons for withdrawing participation defined.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Total participants that withdrew participation in the study.
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy | Overall
Number analyzed (Participants) | 6 | 1 | 7
Participants
  Scheduling conflicts | 1 | 0 | 1
  Health issues | 2 | 0 | 2
  Lack of privacy | 0 | 1 | 1
  Reimbursement issues | 1 | 0 | 1
  Reasons unknown | 2 | 0 | 2

8. Primary Outcome: Feasibility as Assessed by Participants Lost to Follow-Up
Description: Includes the number of individuals who were lost to follow-up and unable to be traced (N=5).
Time Frame: Assessed up to 6 months post-baseline
Population: The "Overall Number of Participants Analyzed" below reflect the number of enrolled participants in each study arm. Participants who were lost to follow-up (n=5) were part of both the intervention arm (n=2) and the control arm (n=3).
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Total participants that were lost to follow-up.
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy | Overall
Number analyzed (Participants) | 23 | 21 | 44
Participants | 2 | 3 | 5

9. Primary Outcome: Acceptability of Study Procedures, as Assessed by the Client Satisfaction Questionnaire
Description: Investigators assessed acceptability at the post-treatment visit using the eight-item Client Satisfaction Questionnaire (CSQ-8), a measure of how much an individual values a treatment. Items are summed to create an overall score; scores range from 8 to 32, with higher scores indicating higher satisfaction. Excellent acceptability was defined a priori as CSQ-8 scores between 26 and 32, and good acceptability was defined a priori as CSQ-8 scores between 20 and 25.
Time Frame: Assessed up to 6 months post-baseline
Population: CSQ-8 scores were collected at the post-treatment assessment; therefore, the "Overall Number of Participants Analyzed" reflects the total number of participants that completed a post-treatment assessment (N=33 overall; N=15 in intervention arm; N=18 in control arm).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy | Overall
Number analyzed (Participants) | 15 | 18 | 33
score on a scale | 20.6 (4.3) | 20.3 (3.5) | 20.4 (3.8)

10. Primary Outcome: Acceptability of Study Procedures, as Assessed by the Perception of Study Assessments Questionnaire
Description: Investigators assessed acceptability at the post-treatment visit by asking participants about their perceptions of the burden of the study assessment battery on a scale from 1 ("no/minimal burden") to 10 ("too much of a burden"). Items are summed to create an overall score; scores range from 1 to 10, with lower scores indicating higher satisfaction.
Time Frame: Assessed up to 6 months post-baseline
Population: Perception of Study Assessment scores were collected at the post-treatment assessment; therefore, the "Overall Number of Participants Analyzed" reflects the total number of participants that completed a post-treatment assessment (N=33 overall; N=15 in intervention arm; N=18 in control arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy | Overall
Number analyzed (Participants) | 15 | 18 | 33
Participants
  "No/minimal burden" (score = 1) | 11 | 9 | 20
  Between "No/minimal burden" and "Moderate burden" (score = 2-4) | 1 | 6 | 7
  Between "Moderate burden" and "Too much of a burden" (score = 5-9) | 2 | 2 | 4
  "Too much of a burden" (score = 10) | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 6 months post-baseline
Arm/Group | Intervention Group: Adapted 3RP | Control Group: Supportive Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group: Adapted 3RP (N=23) | Control Group: Supportive Psychotherapy (N=21)
Admission to Emergency Department, Unrelated to Study (Psychiatric disorders) | 1 (1) | 0 — An enrolled participant who had not attended group sessions was admitted to the Emergency Department for depression. The participant was connected to mental health care. The IRB determined that this SAE was unrelated to the study and not reportable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT03673098/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03673098/ICF_001.pdf